CLINICAL TRIAL: NCT01285323
Title: A 12-Month, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Reslizumab (3.0 mg/kg) in the Reduction of Clinical Asthma Exacerbations in Patients (12-75 Years of Age) With Eosinophilic Asthma
Brief Title: A Study to Evaluate the Efficacy and Safety of Reslizumab in Patients With Eosinophilic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C38072/3083; 2010-024006-35 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-28 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — reslizumab; Antibodies, Monoclonal, Humanized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered intravenously once every 4 weeks ( +-7 days) for a total of 13 doses.
  Interventions: Drug: Placebo
- Reslizumab 3.0 mg/kg (Experimental): Reslizumab 3.0 mg/kg administered intravenously once every 4 weeks ( +-7 days) for a total of 13 doses.
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — Patients were administered intravenously over 15 to 30 minutes reslizumab at a dosage of 3.0 mg/kg at baseline and once every 4 weeks relative to baseline over 48 weeks for a total of 13 doses.
  Other Names: Cinquil; humanized monoclonal antibody; CEP-38072
  Arms: Reslizumab 3.0 mg/kg
Drug: Placebo — Matching placebo (acetate sucrose buffer), administered intravenously (iv) once every 4 weeks for a total of 13 doses.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether reslizumab is more effective than placebo in reducing the number of clinical asthma exacerbations (CAEs) in patients with eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female, 12 through 75 years of age, with a previous diagnosis of asthma. Patients 12 through 17 years of age are excluded from participating in Germany, India, Argentina, and Korea; patients 66 through 75 years of age are excluded from participating in India and Korea.
* The patient has had at least 1 asthma exacerbation requiring oral, intramuscular (im), or intravenous (iv) corticosteroid use for at least 3 days over the past 12 months before screening.
* The patient has a current blood eosinophil level of at least 400/μL.
* The patient has airway reversibility of at least 12% to beta-agonist administration.
* The patient has an ACQ score of at least 1.5 5 at the screening and baseline (before the 1st dose of study drug) visits.
* The patient is taking inhaled fluticasone at a dosage of at least 440 μg, or equivalent, daily. Chronic oral corticosteroid use (no more than 10 mg/day prednisone or equivalent) is allowed. If a patient is on a stable dose, eg, 2 weeks or more of oral corticosteroid treatment at the time of study enrollment, the patient must remain on this dose throughout the study. The patient's baseline asthma therapy regimen (including, but not limited to, inhaled corticosteroids, oral corticosteroids up to a maximum dose of 10 mg prednisone daily or equivalent, leukotriene antagonists, 5-lipoxygenase inhibitors, or cromolyn) must be stable for 30 days prior to screening and baseline and must continue without dosage changes throughout the study.
* All female patients must be surgically sterile, 2 years postmenopausal, or must have a negative pregnancy test (ß-human chorionic gonadotropin [ß-HCG]) at screening (serum) and baseline (urine).
* Female patients of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include barrier method with spermicide, abstinence, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected). NOTE: Partner sterility alone is not acceptable for inclusion in the study.
* Written informed consent is obtained. Patients 12 through 17 years old, where participating, must provide assent.
* The patient is in reasonable health (except for diagnosis of asthma) as judged by the investigator, and as determined by a medical history, medical examination, ECG evaluation (at screening), serum chemistry, hematology, and urinalysis.
* The patient must be willing and able to understand and comply with study restrictions, requirements, and procedures, as specified by the study center, and to remain at the study center for the required duration during the study period, and willing to return to the study center for the follow-up evaluation as specified in this protocol.
* Patients who experience an asthma exacerbation during the screening period will be considered to have failed screening and cannot be randomly assigned to study drug. Patients may be rescreened 1 time only.

Exclusion Criteria:

* The patient has a clinically meaningful co-morbidity that would interfere with the study schedule or procedures, or compromise the patient's safety.
* The patient has known hypereosinophilic syndrome.
* The patient has another confounding underlying lung disorder (eg, chronic obstructive pulmonary disease, pulmonary fibrosis, or lung cancer). Patients with pulmonary conditions with symptoms of asthma and blood eosinophilia (eg, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis) will also be excluded.
* The patient is a current smoker (ie, has smoked within the last 6 months prior to screening).
* The patient is using systemic immunosuppressive, immunomodulating, or other biologic agents (including, but not limited to, anti-immunoglobulin E (IgE) mAb, methotrexate, cyclosporin, interferon-α, or anti-tumor necrosis factor [anti-TNF] mAb) within 6 months prior to screening.
* The patient has previously received an anti-hIL-5 monoclonal antibody (eg, reslizumab, mepolizumab, or benralizumab).
* The patient has any aggravating medical factors that are inadequately controlled (eg, rhinitis, gastroesophageal reflux disease, and uncontrolled diabetes).
* The patient has participated in any investigative drug or device study within 30 days prior to screening.
* The patient has participated in any investigative biologics study within 6 months prior to screening.
* Other exclusion criteria apply.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (104):
- United States (15):
  - Teva Investigational Site 48, Mobile, Alabama
  - Teva Investigational Site 41, Fresno, California
  - Teva Investigational Site 59, Long Beach, California
  - Teva Investigational Site 47, Denver, Colorado
  - Teva Investigational Site 28, Waterbury, Connecticut
  - Teva Investigational Site 53, Clearwater, Florida
  - Teva Investigational Site 27, Miami, Florida
  - Teva Investigational Site 25, Lawrenceville, Georgia
  - Teva Investigational Site 57, Metairie, Louisiana
  - Teva Investigational Site 46, Bangor, Maine
  - Teva Investigational Site 40, St Louis, Missouri
  - Teva Investigational Site 67, Fort Mill, South Carolina
  - Teva Investigational Site 44, Dallas, Texas
  - Teva Investigational Site 69, El Paso, Texas
  - Teva Investigational Site 45, San Antonio, Texas
- Argentina (4):
  - Teva Investigational Site 121, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 126, Ciudad Autonoma de Buenos Aire
  - Teva Investigational Site 123, Rosario-Santa Fe
  - Teva Investigational Site 120, San Miguel de Tucuman - Tucuma
- Brazil (6):
  - Teva Investigational Site 150, Florianópolis
  - Teva Investigational Site 140, Porto Alegre
  - Teva Investigational Site 144, Porto Alegre
  - Teva Investigational Site 145, Porto Alegre
  - Teva Investigational Site 143, Porto Alegre, RS
  - Teva Investigational Site 142, Santo André
- Canada (3):
  - Teva Investigational Site 104, Newmarket
  - Teva Investigational Site 102, Pointe-Claire
  - Teva Investigational Site 105, Windsor
- France (3):
  - Teva Investigational Site 343, Grenoble
  - Teva Investigational Site 342, Marseille
  - Teva Investigational Site 341, Montpellier
- Germany (13):
  - Teva Investigational Site 360, Bad Wörishofen
  - Teva Investigational Site 361, Berlin
  - Teva Investigational Site 362, Berlin
  - Teva Investigational Site 366, Berlin
  - Teva Investigational Site 371, Bochum
  - Teva Investigational Site 365, Dresden
  - Teva Investigational Site 369, Frankfurt
  - Teva Investigational Site 370, Hamburg
  - Teva Investigational Site 372, Koblenz
  - Teva Investigational Site 367, Leipzig
  - Teva Investigational Site 368, Leipzig
  - Teva Investigational Site 363, Mainz
  - Teva Investigational Site 364, Mainz
- Greece (3):
  - Teva Investigational Site 381, Alexandroupoli
  - Teva Investigational Site 380, Athens
  - Teva Investigational Site 382, Heraklion, Crete
- Mexico (6):
  - Teva Investigational Site 203, Distrito Federal
  - Teva Investigational Site 204, Guadalajara, JAL
  - Teva Investigational Site 205, Mexico City
  - Teva Investigational Site 207, Mexico City
  - Teva Investigational Site 209, Monterrey
  - Teva Investigational Site 202, Tijuana, B.C.
- Peru (8):
  - Teva Investigational Site 223, Cercado de Lima, Lima
  - Teva Investigational Site 220, Lima
  - Teva Investigational Site 221, Lima
  - Teva Investigational Site 222, Lima
  - Teva Investigational Site 225, Lima
  - Teva Investigational Site 226, Lima
  - Teva Investigational Site 227, Lima
  - Teva Investigational Site 229, Lima
- Romania (5):
  - Teva Investigational Site 523, Bucharest
  - Teva Investigational Site 524, Bucharest
  - Teva Investigational Site 520, Cluj-Napoca
  - Teva Investigational Site 521, Iași
  - Teva Investigational Site 522, Târgu Mureş
- Russia (9):
  - Teva Investigational Site 543, Moscow
  - Teva Investigational Site 544, Moscow
  - Teva Investigational Site 554, Moscow
  - Teva Investigational Site 556, Moscow
  - Teva Investigational Site 558, Moscow
  - Teva Investigational Site 559, Moscow
  - Teva Investigational Site 557, Novosibirsk
  - Teva Investigational Site 540, Saint Petersburg
  - Teva Investigational Site 541, Saint Petersburg
- Slovakia (4):
  - Teva Investigational Site 563, Bradejov
  - Teva Investigational Site 561, Levice
  - Teva Investigational Site 560, Spišská Nová Ves
  - Teva Investigational Site 562, Topoľčany
- South Korea (6):
  - Teva Investigational Site 682, Gwangju
  - Teva Investigational Site 680, Seoul
  - Teva Investigational Site 681, Seoul
  - Teva Investigational Site 683, Seoul
  - Teva Investigational Site 686, Seoul
  - Teva Investigational Site 685, Suwon
- Taiwan (5):
  - Teva Investigational Site 764, Kaohsiung City
  - Teva Investigational Site 765, Taichung
  - Teva Investigational Site 760, Taipei
  - Teva Investigational Site 761, Taipei
  - Teva Investigational Site 763, Taoyuan District
- Ukraine (14):
  - Teva Investigational Site 621, Dnipropetrovsk
  - Teva Investigational Site 629, Donetsk
  - Teva Investigational Site 635, Donetsk
  - Teva Investigational Site 630, Ivano-Frankivsk
  - Teva Investigational Site 620, Kharkiv
  - Teva Investigational Site 633, Kharkiv
  - Teva Investigational Site 622, Kyiv
  - Teva Investigational Site 623, Kyiv
  - Teva Investigational Site 624, Kyiv
  - Teva Investigational Site 625, Kyiv
  - Teva Investigational Site 628, Ternopil
  - Teva Investigational Site 626, Vinnytsia
  - Teva Investigational Site 631, Zaporizhzhia
  - Teva Investigational Site 632, Zaporizhzhia

REFERENCES:
- [Derived] Nair P, Bardin P, Humbert M, Murphy KR, Hickey L, Garin M, Vanlandingham R, Chanez P. Efficacy of Intravenous Reslizumab in Oral Corticosteroid-Dependent Asthma. J Allergy Clin Immunol Pract. 2020 Feb;8(2):555-564. doi: 10.1016/j.jaip.2019.09.036. Epub 2019 Oct 15. PMID 31626990
- [Derived] Carr WW, McDonald M, Meizlik P. Effect of intravenously administered reslizumab on spirometric lung age in patients with moderate-to-severe eosinophilic asthma. Allergy Asthma Proc. 2019 Jul 1;40(4):240-249. doi: 10.2500/aap.2019.40.4225. PMID 31262379
- [Derived] Han S, Kim S, Kim H, Suh HS. Cost-utility analysis of reslizumab for patients with severe eosinophilic asthma inadequately controlled with high-dose inhaled corticosteroids and long-acting beta2-agonists in South Korea. Curr Med Res Opin. 2019 Sep;35(9):1597-1605. doi: 10.1080/03007995.2019.1605159. Epub 2019 May 16. PMID 30964365
- [Derived] Bateman ED, Djukanovic R, Castro M, Canvin J, Germinaro M, Noble R, Garin M, Buhl R. Predicting Responders to Reslizumab after 16 Weeks of Treatment Using an Algorithm Derived from Clinical Studies of Patients with Severe Eosinophilic Asthma. Am J Respir Crit Care Med. 2019 Feb 15;199(4):489-495. doi: 10.1164/rccm.201708-1668OC. PMID 30346831
- [Derived] Weinstein SF, Katial RK, Bardin P, Korn S, McDonald M, Garin M, Bateman ED, Hoyte FCL, Germinaro M. Effects of Reslizumab on Asthma Outcomes in a Subgroup of Eosinophilic Asthma Patients with Self-Reported Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2019 Feb;7(2):589-596.e3. doi: 10.1016/j.jaip.2018.08.021. Epub 2018 Sep 5. PMID 30193936
- [Derived] Brusselle G, Germinaro M, Weiss S, Zangrilli J. Reslizumab in patients with inadequately controlled late-onset asthma and elevated blood eosinophils. Pulm Pharmacol Ther. 2017 Apr;43:39-45. doi: 10.1016/j.pupt.2017.01.011. Epub 2017 Jan 31. PMID 28159511
- [Derived] Castro M, Zangrilli J, Wechsler ME, Bateman ED, Brusselle GG, Bardin P, Murphy K, Maspero JF, O'Brien C, Korn S. Reslizumab for inadequately controlled asthma with elevated blood eosinophil counts: results from two multicentre, parallel, double-blind, randomised, placebo-controlled, phase 3 trials. Lancet Respir Med. 2015 May;3(5):355-66. doi: 10.1016/S2213-2600(15)00042-9. Epub 2015 Feb 23. PMID 25736990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1111 patients were screened for this study. Of the 1111 patients screened, 464 patients at 82 centers in 15 countries were randomly assigned to double-blind treatment.
Period: Overall Study
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Started | 232 | 232
Full Analysis Set | 232 (Randomized participants who received at least 1 dose of study drug) | 232
Safety Analysis Set | 232 (Participants who received at least 1 dose of study drug) | 232
Completed | 199 | 202
Not Completed | 33 | 30
Not completed — Adverse Event | 9 | 8
Not completed — Lack of Efficacy | 4 | 2
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Protocol Violation | 1 | 2
Not completed — Non-compliance with study procedures | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reslizumab 3.0 mg/kg | Total
Number analyzed (Participants) | 232 | 232 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.75) | 46.4 (13.79) | 47.0 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 144 | 294
  Male | 82 | 88 | 170
Race [Number; unit: participants]
  White | 169 | 168 | 337
  Black | 4 | 6 | 10
  Asian | 21 | 16 | 37
  American Indian or Alaskan Native | 4 | 7 | 11
  Pacific Islander | 1 | 0 | 1
  Other | 33 | 35 | 68
Weight [Mean (Standard Deviation); unit: kg] | 73.9 (15.93) | 74.7 (15.72) | 74.3 (15.81)
Height [Mean (Standard Deviation); unit: cm] | 165.2 (9.81) | 166.4 (9.56) | 165.8 (9.69)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27 (5.05) | 27 (5.26) | 27 (5.15)
Oral Corticosteroid Use at Baseline [Number; unit: participants] — Participants who were taking oral corticosteroids at baseline as recorded by interactive response technology. This was a stratification factor.
  participants
    Yes | 27 | 27 | 54
    No | 205 | 205 | 410
Participants in the United States [Number; unit: participants] — This was a stratification factor as reported by the interactive response technology (IRT).
  participants
    Yes | 15 | 16 | 31
    No | 217 | 216 | 433
Asthma exacerbations in the previous 12 months [Mean (Standard Deviation); unit: exacerbations] — One Reslizumab participant reported no asthma exacerbations in the past 12 months.
  exacerbations | 2.0 (1.78) | 1.9 (1.58) | 1.9 (1.68)
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] | 2.004 (0.6682) | 2.129 (0.7848) | 2.066 (0.7307)
Asthma Control Questionnaire (ACQ) [Mean (Standard Deviation); unit: units on a scale] — The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the overall score is the mean of all responses. A higher score is an indication of poorer asthma control.
  units on a scale | 2.605 (0.79) | 2.570 (0.89) | 2.587 (0.84)
Asthma Quality of Life Questionnaire (AQLQ) [Mean (Standard Deviation); unit: units on a scale] — The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses.
  units on a scale | 4.223 (1.0794) | 4.352 (1.0220) | 4.287 (1.0521)
Asthma Symptom Utility Index (ASUI) [Mean (Standard Deviation); unit: units on a scale] — The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control.
  units on a scale | 0.649 (0.1919) | 0.664 (0.2005) | 0.656 (0.1961)
Blood Eosinophil Count [Mean (Standard Deviation); unit: 10^9 blood eosinophil/L] | 0.688 (0.6824) | 0.610 (0.4115) | 0.649 (0.5642)
Number of Short-Acting Beta-Agonist Puffs (SABA) Daily [Mean (Standard Deviation); unit: puffs/day] — Based on patient-reported total number of SABA puffs over the past 3 days. N=201, 204, 405
  puffs/day | 2.7 (2.41) | 2.9 (2.82) | 2.8 (2.62)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Clinical Asthma Exacerbations (CAEs) During 12 Months of Treatment
Description: An exacerbation event was considered a CAE if the patient met either or both of the criteria listed below and this was corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:
  * use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days; or an increased 2 or more fold for at least 3 or more days for patient's already on corticosteroids.
  * asthma-related emergency treatment, such as an unscheduled visit to the physician's office or emergency room for nebulizer treatment or other urgent treatment to prevent worsening of asthma symptoms, or an asthma-related hospitalization.
  CAEs were adjudicated by committee to assure consistency. Adjusted CAE rate and confidence intervals were based on Negative Binomial regression model adjusted for stratification factors.
  Results are offered as adjusted means.
Time Frame: Day 1 to Month 12
Population: Randomized set includes all patients who were randomly assigned to a treatment group at enrollment, regardless of whether or not a patient took any study drug.
Measure: Mean (95% Confidence Interval); unit: CAEs in 52 weeks
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 232 | 232
CAEs in 52 weeks | 2.115 [1.329 to 3.365] | 0.859 [0.549 to 1.345]
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group and randomization stratification factors as model factors and the logarithm of follow up time excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority or Other; p < 0.0001, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio (reslizumab vs placebo) = 0.4063, 95% CI 2-sided [0.2819 to 0.5855]

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) At Week 16
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma obtained from pulmonary function tests. It is the volume of air expired in the first second of a forced expiration using a spirometer.
  Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Week 16
Population: Randomized set includes all patients who were randomly assigned to a treatment group at enrollment, regardless of whether or not a patient took any study drug. Number analyzed reflects participants with both baseline and Week 16 assessments.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 214 | 214
liters | 0.122 (0.0447) | 0.223 (0.0445)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; A pre-specified fixed sequence multiple testing procedure was implemented to test the secondary endpoints while controlling the overall Type I error rate at 0.05. At the point where p>0.05, no further comparisons were interpreted inferentially; Test type: Superiority or Other; p = 0.0109, Mixed model repeated measures (MMRM) — Statistical significance at <=0.05; Fixed Factors: treatment, visit, trt by visit interaction, region, OCS at enrollment, sex. Random: covariates for height, baseline value and patient; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.023 to 0.179], Standard Error of Mean 0.0397 — active - placebo

3. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: FEV1 is a standard measurement of air movement in the lungs of patients with asthma obtained from pulmonary function tests. It is the volume of air expired in the first second of a forced expiration using a spirometer. During study (Weeks 4, 8, 12 and 16) average value used a mixed effect model for repeated measures (MMRM) with treatment group, visit, treatment and visit interaction, and stratification factors as fixed effects and participant as a random effect. Covariates for baseline values were also included in the model; for pulmonary function test analyses, covariates for height and sex were included as well.
  Positive change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12 and 16
Population: Randomized set includes all patients who were randomly assigned to a treatment group at enrollment, regardless of whether or not a patient took any study drug. Includes participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 227 | 230
liters | 0.094 (0.041) | 0.187 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0037, Mixed model repeated measures (MMRM) — Statistical significance at <=0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [0.030 to 0.155], Standard Error of Mean 0.0317 — active-placebo

4. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) to Week 16
Description: The AQLQ is a 32-item instrument administered as a self-assessment (Juniper et al 1992). The questionnaire is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Patients were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (1=severe impairment, 7=no impairment). The overall AQLQ score is the mean of all 32 responses. Five of the activity questions were "patient-specific," which means that each patient identified and scored 5 activities in which the patient was limited by asthma; these 5 activities were identified at the first visit and retained for all subsequent follow-up visits.
  Positive change from baseline scores indicate improvement in quality of life.
Time Frame: Day 1 (baseline, pre-dose), Week 16
Population: Randomized set of participants with assessments at each timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 216 | 213
units on a scale | 0.777 (0.1152) | 0.987 (0.1158)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0259, Mixed model repeated measures (MMRM) — Statistical significance at <=0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.209, 95% CI 2-sided [0.025 to 0.393], Standard Error of Mean 0.937 — active - placebo

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ACQ is a 7-item instrument that measures asthma control (Juniper et al 1999). Six questions are self-assessments; the seventh item, completed by a member of the study staff, is the result of the patient's FEV1 measurement. Each item has 7 possible answers on a scale of 0 to 6, and the total score is the mean of all responses (the total scale is therefore 0-6). A higher score is an indication of poorer asthma control. The during treatment (Weeks 4, 8, 12 and 16) average ACQ was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Randomized set, including participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 228 | 230
units on a scale | -0.660 (0.0875) | -0.857 (0.0872)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0032, Mixed model repeated measures (MMRM) — Statistical significance at <=0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.196, 95% CI 2-sided [-0.327 to -0.066], Standard Error of Mean 0.0664 — active - placebo

6. Secondary Outcome: Kaplan-Meier Estimates for Time to First Clinical Asthma Exacerbation (CAE)
Description: An exacerbation event was considered a CAE if the patient met either or both of the criteria listed below and this was corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:
  * use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days; or an increased 2 or more fold for at least 3 or more days for patient's already on corticosteroids.
  * asthma-related emergency treatment, such as an unscheduled visit to the physician's office or emergency room for nebulizer treatment or other urgent treatment to prevent worsening of asthma symptoms, or an asthma-related hospitalization.
  CAEs were adjudicated by committee to assure consistency. The distributions were compared by a log rank test stratified by baseline usage of oral corticosteroid (yes or no) and geographical region (US or other).
Time Frame: Day 1 to Day 526 (longest treatment time plus 2 weeks)
Population: Randomized set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 232 | 232
weeks | NA [NA to NA] — Insufficient data to estimate time | NA [NA to NA] — Insufficient data to estimate time
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; Kaplan-Meier estimate of probability (5) of not experiencing a CAE by week 52. The first CAEs for each patient occurring after randomization and up to 2 weeks after the end of treatment period were analyzed. Patients without a CAE within this time frame were censored at two weeks after the treatment completion date or study discontinuation, whichever came first; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Stratified by baseline usage of oral corticosteroid (yes or no) and geographical region (US or other); Hazard Ratio (HR) = 0.486, 95% CI 2-sided [0.353 to 0.670] — Reslizumab vs placebo

7. Secondary Outcome: Change From Baseline in Asthma Symptom Utility Index (ASUI) Over 16 Weeks Using Mixed Model for Repeated Measures
Description: The ASUI is an 11-item instrument designed to assess the frequency and severity of asthma symptoms and side effects, weighted by patient preferences (Revicki et al 1998). ASUI is a utility score that ranges from 0 to 1, with higher values indicating better asthma control; info obtained from questionnaire about asthma symptoms.
  The during treatment (Weeks 4, 8, 12 and 16) average ASUI was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Positive change from baseline values indicate improvement in asthma symptoms. Information was obtained from questionnaire about asthma symptoms.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Randomized set, including participants who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 224 | 227
units on a scale | 0.080 (0.0161) | 0.115 (0.0161)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0037, Mixed model repeated measures (MMRM) — Statistical significance at <=0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [0.011 to 0.059], Standard Error of Mean 0.0120 — active - placebo

8. Secondary Outcome: Change From Baseline in Short-Acting Beta-Agonist (SABA) Use Over 16 Weeks Using Mixed Model for Repeated Measures
Description: SABA are used for quick relief of asthma symptoms. To measure SABA use, at each clinical visit patients were asked to recall their usage of SABA therapy within the last 3 days of the scheduled visit. If usage was confirmed, the number of puffs used was recorded. For the purpose of summaries, an average daily usage was evaluated by dividing the total number of puffs recorded over 3 days by 3.
  The during treatment (Weeks 4, 8, 12 and 16) average SABA use was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements.
  Negative change from baseline scores indicate improvement in asthma control.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16
Population: Randomized set including patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: SABA puffs per day
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 188 | 180
SABA puffs per day | -0.44 (0.233) | -0.50 (0.230)
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7263, Mixed model repeated measures (MMRM) — Statistical significance at <=0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.062, 95% CI 2-sided [-0.411 to 0.287], Standard Error of Mean 0.1775 — active - placebo

9. Secondary Outcome: Change From Baseline in Blood Eosinophil Count Over 16 Weeks and 52 Weeks Using Mixed Model for Repeated Measures
Description: The blood eosinophil counts were measured using a standard complete blood count (CBC) with differential blood test. Results of all differential blood tests conducted after randomization were blinded.
  The during treatment average eosinophil count was estimated using a mixed-effect model for repeated measures (MMRM) with fixed effects (treatment, stratification factors, sex, visit, interaction of treatment and visit), covariates (height, baseline value), and patient as the random effect for the repeated measurements. The 'over 16 weeks' value used data from Weeks 4, 8, 12 and 16. The 'over 52 weeks' value used all the during study time points listed in the Time Frame field.
  Negative change from baseline values correlate to reduced asthma severity.
Time Frame: Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 or early withdrawal
Population: Randomized set including patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: 10^9 blood eosinophil/L
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 226 | 230
10^9 blood eosinophil/L
  Over first 16 weeks | -0.076 (0.0268) | -0.555 (0.0266)
  Over 52 weeks | -0.076 (0.0233) | -0.565 (0.0231)

10. Secondary Outcome: Participants With Treatment-Emergent Adverse Events TEAE)
Description: An adverse event (AE) was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 (post-dose) to Week 65. The endpoint for adverse events was the last postbaseline observation, which included the 90 day follow-up visit.
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 232 | 232
participants
  Any TEAE | 201 | 177
  Mild TEAE | 36 | 67
  Moderate TEAE | 140 | 98
  Severe TEAE | 25 | 12
  Treatment-related AE | 27 | 34
  Mild treatment-related AE | 14 | 22
  Moderate treatment-related AE | 13 | 11
  Severe treatment-related AE | 0 | 1
  TEAE causing patient discontinuation | 9 | 8
  Deaths | 0 | 0
  Serious AEs | 23 | 18

11. Primary Outcome: Frequency of Each of the Two Criteria for Clinical Asthma Exacerbations (CAEs)
Description: An exacerbation event was considered a CAE if the patient met either or both of the criteria listed below and this was corroborated with at least 1 other measurement to indicate the worsening of clinical signs and symptoms of asthma:
  * use of systemic, or an increase in the use of inhaled, corticosteroid treatment for 3 or more days; or an increased 2 or more fold for at least 3 or more days for patient's already on corticosteroids.
  * asthma-related emergency treatment, such as an unscheduled visit to the physician's office or emergency room for nebulizer treatment or other urgent treatment to prevent worsening of asthma symptoms, or an asthma-related hospitalization CAEs were adjudicated by committee to assure consistency.
  Adjusted CAE rate and confidence intervals for the two criteria were based on Negative Binomial regression model adjusted for stratification factors.
  Results are offered as adjusted means.
Time Frame: Day 1 to Month 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: CAEs in 52 weeks
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 232 | 232
CAEs in 52 weeks
  Requiring systemic corticosterioids >3 days | 1.660 [1.005 to 2.744] | 0.646 [0.397 to 1.053]
  Requiring hospitalization or ER visit | 0.047 [0.013 to 0.168] | 0.033 [0.009 to 0.120]
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 3.0 mg/kg; CAE Due to Requiring Systemic Corticosteroids The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group and randomization stratification factors as model factors and the logarithm of follow up time excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority or Other; p < 0.0001, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio (reslizumab vs placebo) = 0.3893, 95% CI 2-sided [0.2621 to 0.5782]
Statistical Analysis 2: Comparison: Placebo vs Reslizumab 3.0 mg/kg; CAE Due to Hospitalization or ER visit The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group and randomization stratification factors as model factors and the logarithm of follow up time excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority or Other; p = 0.4020, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio = 0.6686, 95% CI 2-sided [0.2878 to 1.6479]

12. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Abnormal Lab Values
Description: Data represents participants with potentially clinically significant (PCS) abnormal serum chemistry, hematology (except for eosinophil values), and urinalysis values.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Creatinine: >=177 μmol/L
  * Urate: M>=625, F>=506 μmol/L
  * Aspartate aminotransferase (AST): >=3*upper limit of normal (ULN)
  * Alanine aminotransferase (ALT): >=3*ULN
  * GGT = gamma-glutamyl transpeptidase: >= 3*ULN
  * Total bilirubin: >=34.2 μmol/L
  * White blood cells (low): <=3.0*10^9/L
  * White blood cells (high): >=20*10^9/L
  * Hemoglobin (age >=18 years): M<=115, F<=95 g/dL
  * Hematocrit (age >=18 years): M<0.37, F<0.32 L/L
  * Eosinophils/leukocytes: >=10.0%
  * Platelets: <=75*10^9/L
  * Neutrophils: <=1.0*10^9/L
  * Urinalysis: blood, ketones, glucose, and protein: >=2 unit increase from baseline
Time Frame: Week 4 to Week 52
Population: Safety analysis set, including participants who contributed to the analysis
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 227 | 230
participants
  Blood urea nitrogen | 5 | 4
  Creatinine | 0 | 1
  Urate | 5 | 2
  AST | 3 | 2
  ALT | 7 | 3
  GGT | 11 | 9
  Bilirubin | 3 | 3
  Leukocytes (low) | 3 | 10
  Leukocytes (high) | 0 | 1
  Hemoglobin | 5 | 6
  Hematocrit | 10 | 8
  Eosinophils/leukocytes | 168 | 10
  Platelets | 1 | 1
  Neutrophils | 14 | 9
  Urine blood (hemoglobin) | 28 | 12
  Urine ketones | 6 | 1
  Urine glucose | 9 | 7
  Urine protein | 28 | 28

13. Secondary Outcome: Participants With Treatment-Emergent Potentially Clinically Significant (PCS) Vital Signs Values
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Sitting pulse (high): >100 and increase of >= 30 beats/minute
  * Sitting systolic blood pressure (low): <90 and decrease of >= 30 mmHg
  * Sitting systolic blood pressure (high): >160 and increase of >= 30 mmHg
  * Sitting diastolic blood pressure (low): <50 and decrease of >=12 mmHg (if 12-17 years old: <55 and decrease of >=12 mmHg 0
  * Sitting diastolic blood pressure (high): >100 and increase of >=12 mmHg
  * Respiratory rate (low): <6 breaths/minute
  * Respiratory rate (high): >24 and increase of >=10 breaths/minute
  * Body temperature (low): <35.8° Celsius
  * Body temperature (high): >=38.1 and increase of >=1.1° Celsius
Time Frame: Week 4 to Week 52
Population: Safety analysis set including participants who contributed data to the analysis
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 230 | 230
participants
  >=1 postbaseline vital sign abnormality | 58 | 49
  Sitting pulse (high) | 6 | 6
  Sitting systolic blood pressure (low) | 2 | 1
  Sitting systolic blood pressure (high) | 0 | 1
  Sitting diastolic blood pressure (low) | 4 | 3
  Sitting diastolic blood pressure (high) | 3 | 4
  Respiratory rate (low) | 0 | 1
  Respiratory rate (high) | 4 | 5
  Body temperature (low) | 50 | 39
  Body temperature (high) | 1 | 0

14. Secondary Outcome: Participants With a Positive Anti-Reslizumab Antibody Status During Study
Description: Counts of participants with a positive anti-drug antibody (ADA) response during treatment is offered for the experimental treatment arm. Blood samples were collected for determination of ADAs before study drug infusion.
Time Frame: Baseline visit (prior to reslizumab exposure), Weeks 16, 32, 48 and 52
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Number analyzed (Participants) | 0 | 232
participants
  Baseline |  | 10
  Week 16 |  | 10
  Week 32 |  | 10
  Week 48 |  | 10
  Week 52 |  | 10
  >=1 positive test result |  | 15

ADVERSE EVENTS:
Time Frame: Day 1 (post-dose) to Week 65. The endpoint for adverse events was the last postbaseline observation, which included the 90 day follow-up visit.
Arm/Group | Placebo | Reslizumab 3.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 23/232 | 18/232
Other Adverse Events (participants affected / at risk) | 160/232 | 123/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=232) | Reslizumab 3.0 mg/kg (N=232)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium fortuitum infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=232) | Reslizumab 3.0 mg/kg (N=232)
Bronchitis (Infections and infestations) | 14 (15) | 2 (5)
Nasopharyngitis (Infections and infestations) | 56 (88) | 45 (71)
Upper respiratory tract infection (Infections and infestations) | 16 (27) | 8 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 12 (13)
Headache (Nervous system disorders) | 16 (20) | 33 (55)
Asthma (Respiratory, thoracic and mediastinal disorders) | 118 (293) | 66 (133)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.